CLINICAL TRIAL: NCT03488901
Title: Prediction of Chemoresistance in Patients Treated for Gestational Trophoblastic Tumors
Brief Title: Chemoresistance of Trophoblastic Tumors
Acronym: PrediCTTro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_807
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Trophoblastic Tumor
MeSH Terms: conditions — Trophoblastic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin fixed and paraffin embedded tissue samples of gestational choriocarcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- methotrexate sensitive: patients with gestational choriocarcinoma cured with methotrexate alone
  Interventions: Other: chemoresistance signature
- methotrexate resistant: patients with gestational choriocarcinoma not cured with methotrexate alone
  Interventions: Other: chemoresistance signature
- polychemotherapy sensitive: patients with gestational choriocarcinoma cured with polychemotherapy
  Interventions: Other: chemoresistance signature
- polychemotherapy resistant: patients with gestational choriocarcinoma not cured with polychemotherapy
  Interventions: Other: chemoresistance signature
- hydatidiform moles without malignant transformation: patients treated for hydatidiform moles but who did not turn into trophoblastic tumors (=controls)
  Interventions: Other: chemoresistance signature
- placental site trophoblastic tumors: patients with placental site trophoblastic tumors not cured with polychemotherapy
  Interventions: Other: chemoresistance signature

INTERVENTIONS:
Other: chemoresistance signature — to study the predictive value of a tissue transcriptomic profile (=chemoresistance signature) in the chemoresistance to single or multiagent chemotherapy

SUMMARY:
Gestational trophoblastic tumors are characterized by their development from placental tissue and their high invasive and metastatic potential. These are rare tumors (1/50 000 pregnancies) affecting young women for whom conservative fertility treatments are preferred. The therapeutic strategy is based on a chemotherapy whose choice of protocol is based on a clinico-biological score, FIGO score, which includes tumor size, gonadotropic chorionic hormone level used as quantitative tumor marker, number and localization. metastases. A FIGO score ≤6 allows the use of monochemotherapy (methotrexate) with a 5-year survival of approximately 99.7%. Scores of 7 to 12 and ≥13 require multidrug therapy (EMA-CO) and are associated with 5-year survival of 95.1% and 61.6%, respectively.

The chemotherapies currently used for the treatment of trophoblastic tumors have been described between the 1950s (methotrexate) and the 1980s (EMA-CO) and have a well documented toxicity regarding the risk of secondary tumors, early menopause or even death by toxicity. .

To date, apart from the FIGO score, there is no predictor of resistance to chemotherapy in gestational trophoblastic tumors. However, among patients with a FIGO score ≤6 and receiving methotrexate in the first line, 9 to 46% will have a resistance and require a second line of treatment. Similarly, if the score is ≥7, 10 to 30% of patients receiving EMA-CO will require at least a second line of multidrug therapy.

The hypothesis of PrediCTTro study is that tissue samples of gestational choriocarcinoma present a transcriptomic profile associated with the risk of further resistance to single or multiagent chemotherapy.

The objective of PrediCTTro is to identify a transcriptomic signature able to predict resistance to single or multiagent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* confirmed gestational trophoblastic tumor histology
* hCG follow-up of at least 12 months after hCG normalization
* registration in the French Reference Center for Trophoblastic Diseases

Exclusion Criteria:

* tissue specimen (block/biopsy) not available
* degraded quality of tissue sample not compatible with transcriptome analysis (>20% of necrosis)

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Patients diagnosed with gestational trophoblastic tumors
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Transcription profile associated with the resistance to chemotherapy | 10 months
  The expression level of 800 genes involved in oncogenesis canonical pathways and immune tolerance will be assessed and correlated with the resistance to single or multiagent chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Français de Référence des Maladies Trophoblastiques, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No